CLINICAL TRIAL: NCT05081661
Title: The Effects of Mental Imagery on Postural Control Following Anterior Cruciate Ligament Plasty - a Pilot Study of Feasibility
Brief Title: Effects of Corporal Visualisation Program of the Static and Dynamic Balance After an Operation of the LCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HES-SO Valais-Wallis (Other)
Responsible Party: Principal Investigator, Marielle Pirlet, MSc Physiotherapist - Senior lecturer, HES-SO Valais-Wallis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IM - CP - LCA
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: ACL plasty; anterior cruciate ligament; motor imagery; postural control
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Imagery Group A (Experimental): This group will follow a program of motor imagery.
  Interventions: Other: Motor Imagery Program
- Motor Imagery Group B (Placebo Comparator): This group will follow a placebo program inspired from Bodyscan
  Interventions: Other: Placebo program

INTERVENTIONS:
Other: Motor Imagery Program — The intervention group of the study will undergo standard postoperative physical therapy treatment at their therapist. Beginning on the third day after surgery, the participant will begin an motor imagery program to be performed three times a week for four weeks. A session lasts between fifteen and twenty minutes. It begins with a body awareness phase followed by a series of three to five one-minute exercises to be repeated three times, with a one-minute break between each exercise. The program is performed independently at home using a standardized audio tape.
  Arms: Motor Imagery Group A
Other: Placebo program — The control group of the study will undergo standard postoperative physiotherapy treatment at their therapist. On the third day after surgery, the participant will begin a relaxation program inspired by the mindfulness tool called Bodyscan that acts as a placebo mental imagery program. Nevertheless, the program created for this technique does not follow the Bodyscan guidelines (Jon Kabat-Zinn, 2005), as we do not want there to be any effects in favor of improved body perception on the participants, which could bring an additional biai to the study. For the sake of understanding, we have used the term "body visualization" in the various documents distributed to the participants. The program is to be performed three times a week for four weeks. A session lasts between ten and fifteen minutes. The program is performed independently at home using a standardized audio tape.
  Arms: Motor Imagery Group B

SUMMARY:
The aim of this pilot study is to assess the feasibility of a RCT whose topic would be the effect of a motor imagery program on the postural control in persons who have undergone ACL plasty.

DETAILED DESCRIPTION:
Primary and secondary outcomes will be measured twice at the hospital, a first time six weeks after the beginning of the intervention and a second time eight weeks after the four weeks of the intervention.

Twelves home-based motor imagery sessions will occur in four weeks, three times a week, to activate. The training sessions will last between 15 and 20 minutes. During each training session, the participant will note on his/her own "Tracking sheet" how long they listened to the audio and their comments. The "Tracking sheet" will document whether or not the patient has participated in each of the twelve sessions.

In parallel, a control group will follow a placebo programme according to the same formalities.

Twenty-three participants (min.) will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* men and women of legal age
* to be capable of discernment
* to have a telephone number or email address to communicate with the investigators, to have a device with internet access to access the mental imagery programs.
* to have had an ACL surgery performed by the Doctor Siegrist within the last three days using the Hamstrings Tendon Graft or the Kenneth Jones method.

Exclusion Criteria:

* not having a good spoken knowledge of the French language
* recurrence of ACL injury in the same knee
* meniscal sutures
* associated fractures
* pre-existing balance problems (tested at recruitment)
* pre-existing neurological problems diagnosed by a doctor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 26 Weeks
  Fulfilled if the recruitment rate is above 50% of eligible patients per month.
Enrolment rate | 38 Weeks
  Fulfilled if the participation rate is > 75% (Percentage of participants who completed the study and the full programme, i.e. a minimum of eleven sessions out of twelve)

SECONDARY OUTCOMES:
Dynamic postural control | 12 Weeks
  Modified Star Excursion Balance Test (SEBT), average length in percent
Static postural control | 12 Weeks
  Balance Error Scoring System (BESS), scoring ranges from 0 (best) to 60 (worse
Changes in the functional capacities of the operated knee | 12 Weeks
  Lysholm Questionnaire, Score range from 0 (worse disability) to 100 (less disability)
Mental representation ability | 6 Weeks
  Kinesthetic and Visual Imagery Questionnaire (KVIQ-10), scoring ranges from 0 (worse) to 50 (best)
Use of Electrotherapy | 6 Weeks
  Use of Electrotherapy during the rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Pirlet, master, Principal Investigator — HES-SO Valais-Wallis
Locations (1):
- Marielle.Pirlet, Sion, Switzerland

IPD SHARING:
Plan to Share IPD: No